CLINICAL TRIAL: NCT00693251
Title: Phase IV Study of Optimal Stenting Strategy For True Bifurcation Lesions
Brief Title: Optimal Stenting Strategy For True Bifurcation Lesions
Acronym: PERFECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-0714
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
Keywords: stent; bifurcation; coronary artery stenosis; balloon angioplasty
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Sirolimus; Paclitaxel; zotarolimus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bifurcation stent technique (Experimental): crush technique
  Interventions: Procedure: Crush technique
- bifurcation stent techniqe (Active Comparator): provisional T stenting
  Interventions: Procedure: provisional T stenting

INTERVENTIONS:
Procedure: Crush technique — Crush technique
  Other Names: Sirolimus, Paclitaxel, Zotarolimus and Everolimus stents
  Arms: bifurcation stent technique
Procedure: provisional T stenting — Provisional T stenting
  Other Names: Sirolimus, Paclitaxel, Zotarolimus and Everolimus stents
  Arms: bifurcation stent techniqe

SUMMARY:
It is unclear which stenting strategy will be optimal for true bifurcation coronary lesions.

DETAILED DESCRIPTION:
The outcome of percutaneous coronary intervention of bifurcation lesions with bare-metal stents is hindered by increased rates of procedural complications and long-term major adverse cardiac events compared with non-bifurcated lesions.1 Randomized studies have demonstrated that drug-eluting stents reduce restenosis when used in relatively simple lesions; and recent data have demonstrated efficacy of the sirolimus-eluting stent for bifurcation lesions compared with historical data of BMS. In one study of bifurcation lesions, the overall restenosis rate was 23%, with the majority of side branch restenoses occurring at the ostium after use of a T-stenting technique. Indeed, side branch restenosis occurred in 16.7% after T-stenting, compared with 7.1% after other stenting techniques.

The "crush" technique of bifurcation stenting with DESs was introduced by Colombo et al. in 2003 as a relatively simple technique that ensures complete coverage of the side branch ostium, thereby facilitating drug delivery at this site. Initial data of 20 patients treated with this technique with SES suggest that it is a safe method, with an acceptable rate of procedural complications and no further adverse events up to 30 days follow-up. Recently, angiographic data have shown the importance of simultaneous kissing balloon post-dilation in reducing restenosis and need for target lesion revascularization. They also reported that compared to T-stenting, crushing with final kissing balloon dilatation was associated with lower rate of restenosis and target lesion revascularization. Consequently, the crushing is currently most promising technique in treating bifurcation lesions using two stents. However, despite the advance of bifurcation stenting technique, the superiority of bifurcation stenting with crushing technique over simple stenting in bifurcation lesion has not been demonstrated.

Therefore, we conducted the prospective randomized study comparing crushing technique with final kissing balloon dilatation and a simple technique (main vessel stenting and provisional T-stenting) for treatment of true bifurcation lesions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical

  * Patients with angina and documented ischemia or patients with documented silent ischemia
  * Patients who are eligible for intracoronary stenting
  * Age >18 years, <75 ages
* Angiographic

  * De novo lesion located in a major bifurcation point with the MEDINA classification type 1.1.0, 1.0.0, or 0.1.0
  * Main vessel : >= 2.5 mm in vessel size, >= 50% in diameter stenosis and =< 50 mm in lesion length by visual estimation, in which the lesion seems to be covered with =< 2 stents
  * Side branch : >= 2.0 mm in vessel size, >= 50% in diameter stenosis, and < 20 mm in lesion length by visual estimation, in which the lesion seems to be covered with single stent

Exclusion Criteria:

* History of bleeding diathesis or coagulopathy
* Pregnant
* Known hypersensitivity or contra-indication to contrast agent, heparin, sirolimus and paclitaxel
* Limited life-expectancy (less than 1 year) due to combined serious disease
* ST-elevation acute myocardial infarction < 2 weeks
* Characteristics of lesion:

  * Left main disease
  * In-stent restenosis
  * Graft vessels
  * Chronic total occlusion
  * TIMI flow =< grade 2 in the side branch
* Renal dysfunction, creatinine >= 2.0mg/dL
* Contraindication to aspirin, clopidogrel or cilostazol
* LV ejection fraction =< 35%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2008-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Angiographic binary restenosis rate (diameter stenosis >= 50%) at 8 months in either main or side branch | 8 months

SECONDARY OUTCOMES:
Composite of major cardiac adverse events (MACE) including death, MI, stent thrombosis and ischemia-driven target vessel revascularization | 2 years
Reocclusion rate at the side branch at 8 month angiographic follow-up | 8 months
Late loss at the main vessel and the side branch | 8 months
Restenosis rate at the main vessel and/or side branch | 8 months
Influence of bifurcation angle | 8 months
Influence of new three segment bifurcation QCA software | 8 months
Fluoroscopic time | baseline
Procedure time | baseline
Amount of contrast agent | baseline
Number of used stents | baseline
FFR assessment in the side branch | baseline and 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (12):
- South Korea (12):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Busan Saint Mary's Hospital, Busan
  - Cheongju Saint Mary's Hospital, Cheongju-si
  - Kangwon University Hospital, Chuncheon
  - Chungnam National University Hospital, Daejeon
  - Kyungsang University Hospital, Jinju
  - Hallym University Sacred Heart Hospital, Pyeongchon
  - Catholic University, Kangnam St. Mary's Hospital, Seoul
  - Hallym University Sacred Heart Hospital, Seoul
  - Korea Veterans Hospital, Seoul
  - Aju University Hospital, Suwon
  - Ulsan University Hospital, Ulsan